CLINICAL TRIAL: NCT00399451
Title: Preliminary Study on Submucous Sclerosis of Pharynges With 1% Polidocanol to Treat Obstructive Sleep Apnea (OSA) & Snoring Subjects (SS)
Brief Title: Polidocanol Sclerotherapy of Pharynges for Obstructive Sleep Apnea (OSA) and Snoring Subjects(SS)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liaoyang Central Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYZXYY06002; ACTRNO12606000444583
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2006-11-22 (Estimated); Status verified 2006-11

CONDITIONS: Apnea; Snoring
Keywords: Sleep Apnea,Obstructive; apnea-hypopnea index (AHI); polidocanol; sclerotherapy; pharynges
MeSH Terms: conditions — Apnea; Snoring; Sleep Apnea, Obstructive

INTERVENTIONS:
Drug: Polidocanol Sclerotherapy

SUMMARY:
The aim of this prospective study is to evaluate the results of polidocanol sclerotherapy of pharynx for OSAS & SS,to reduce pharyngeal compliance.

DETAILED DESCRIPTION:
Polidocanol submucous sclerosis in the part of pharynges with 1% polidocanol injection.The injection should be in the retropharyngeal submucosa and lateral pharyngeal bands and lateral pharyngeal submucosa and in front submucosa of soft palate.The injection is multi-point,and each point injection is 0.3~0.5ml;the total quantity/each time is not more than 5ml.Every patient have to be treated about 1~2 time.

ELIGIBILITY:
Inclusion Criteria:

* OSAS & SS which palatopharyngeal collapse.

Exclusion Criteria:

* obstructive sleep apnea syndrome (osas) & snoring subjects (ss),which anatomic narrow result in.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-12; Study Completion 2009-06

PRIMARY OUTCOMES:
apnea-hypopnea index (AHI)is on polysomnography(PSG),to compare AHIanterior and posterior treatment.

SECONDARY OUTCOMES:
Arterial oxygen saturation (SaO2) and body mass index (BMI)will be measured on polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: Youliang YIN, MB, Study Director